CLINICAL TRIAL: NCT01236404
Title: Phase 1/2a, Randomized, Double-Blind Placebo-Controlled, Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Response of PB1023 Injection Following Single and Multiple Ascending Subcutaneous Doses in Adult Subjects With Type 2 Diabetes Mellitus (T2DM)
Brief Title: Phase 1/2a, Randomized, Double-Blind, Placebo-Controlled, Study to Assess Safety, Tolerability, PK and PD Response of PB1023 Injection Following Single and Multiple SQ Doses in Adults With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PhaseBio Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB1023-PT-CL-0001
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PB1023 Injection (Experimental): Subcutaneous injection PB1023
  Interventions: Drug: Single Subcutaneous Dose (Part A) of PB1023 or Placebo (0.9% NaCl); Drug: Multiple (Four Weekly) Subcutaneous Injections (Part B) of PB1023 or Placebo (0.9% NaCl)
- Placebo (0.9% Sodium Chloride Injection) (Placebo Comparator): Subcutaneous Injection Placebo
  Interventions: Drug: Single Subcutaneous Dose (Part A) of PB1023 or Placebo (0.9% NaCl); Drug: Multiple (Four Weekly) Subcutaneous Injections (Part B) of PB1023 or Placebo (0.9% NaCl)

INTERVENTIONS:
Drug: Single Subcutaneous Dose (Part A) of PB1023 or Placebo (0.9% NaCl)
Drug: Multiple (Four Weekly) Subcutaneous Injections (Part B) of PB1023 or Placebo (0.9% NaCl) — Once weekly injections for up to four weeks

SUMMARY:
Primary objective:

To evaluate the safety and tolerability of single and multiple ascending doses of PB1023 administered as a subcutaneous (SC) injection in adult subjects with T2DM.

Secondary objectives:

1. To characterize the pharmacokinetic profile of PB1023 after single and multiple ascending doses of PB1023.
2. To assess the pharmacodynamic response of various single and multiple doses of PB1023 (daily fasting plasma glucose, and serial glucose, c-peptide and insulin levels in response to a liquid Mixed Meal Tolerance Test (MMTT).

ELIGIBILITY:
Inclusion Criteria:

* Males or post menopausal or surgically sterile females age 18-75 years of age inclusive.
* Diagnosed with T2DM for > or = 6 months with HbA1c > or = 6.0% but < or = 9.0% while taking stable doses of one oral antihyperglycemic agent but < or = 8.5% when taking two oral antihyperglycemic agents for up to a maximum of 3 months prior to screening.
* Fasting Plasma glucose between 115 mg/dL and 269 mg/dL.
* Fasting C-peptide of > or = 0.8 ng/mL.
* BMI < or = 40 kg/m2.
* Otherwise stable health except for T2DM.

Exclusion Criteria:

* Currently taking a non-oral antihyperglycemic agent.
* Have taken a PPARg agonist within 90 days of screening.
* Known allergy to an approved or investigational GLP-1 receptor analog/agonist.
* Unstable cardiovascular disease as defined in clinical protocol.
* History, symptoms or signs of pancreatitis or severe gastrointestinal disease.
* Personal or family history of medullary thyroid tumors history of Multiple Endocrine Neoplasia Syndrome Type 2.
* Poor glucose control as defined in clinical protocol.
* Clinically significant renal and/or hepatic dysfunction as defined in clinical protocol.
* Absolute requirement for corticosteroids or received systemic steroids within 90 days prior to PB1023 administration.
* Pregnant or lactating females.
* Known history or active alcohol or drug abuse within 12 months prior to screening.
* Positive for HIV, Hepatitis B surface antigen or Hepatitis C antibodies.
* Participating in any other study within 30 days prior to screening.
* Other medical or psychiatric condition which in the opinion of the investigator would place the subject at increased risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Safety/Tolerability | Screening to Final Visit (up to approximately 10 weeks for SAD and 14 weeks for MAD)
  Safety will be evaluated by analyses of incidence of adverse events of interest (possibly related to the class of drug) and other adverse events. Vital signs, ECGs and safety laboratory parameters will also be presented.

SECONDARY OUTCOMES:
Pharmacokinetic Profile | SAD: Pre-dose, 1, 4, 8, and 12 hours post-dose and Day 1, 2, 3, 5, 7, 10, 14, 21 and 28. MAD: Pre-dose, 1, 4, 8, and 12 hours post-dose and Day 1, 2, 3, 5, pre-dose Days 7, 14 and 21 and at 1, 4, 8, and 12 hours post-dose and Day 22, 23, 26, 28, 35, 42,
  To characterize the PK profile of PB1023 after single and multiple ascending doses of PB1023. The following parameters will be evaluated: t1/2, AUC(inf), AUC(0-t), Tmax, Cmax, Elimination Rate Constant, Clearance and Distribution.
Pharmacodynamic Response | Fasting plasma glucose collected the day before dosing and with PK samples, excluding day of dosing. SAD MMTT to occur on day 0 and 2, MAD MMTT to occur on Day 0 and 22 with continuous glucose monitoring on Day -8/-7 to Day 0 and on Day 21 to Day 28.
  To assess the pharmacodynamic response of various single and multiple doses of PB1023 (daily fasting plasma glucose and serial glucose (and continuous monitoring as defined in time frame), c-peptide and insulin levels in response to a liquid mixed meal tolerance test (MMTT) pre and post dose) on subjects washed off their baseline oral antihyperglycemic agents.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Matson, M.D., Principal Investigator — Prism Research
Locations (3):
- United States (3):
  - Diablo Clinical Research, Walnut Creek, California
  - Prism Research, Saint Paul, Minnesota
  - Rainier Clinical Research Center, Inc., Renton, Washington